CLINICAL TRIAL: NCT03664375
Title: Impact Of Physiotherapy And Botulinum Toxin Type-A In Improving Functional Outcomes In Upper Limb Focal Dystonia Among Post Stroke Patients
Brief Title: Impact Of Physiotherapy And Botox In Improving Functional Outcomes Among Post Stroke Focal Dystonia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Muhammad Umar, Principal Investigator, Isra University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIRS-IUISB/PHD/008
Record Dates: First submitted 2018-09-05; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Focal Hand Dystonia
Keywords: Dystonia Task-specific training Botulinum toxin type A
MeSH Terms: conditions — Dystonia, Focal, Task-Specific | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: A total of 46 patients were recruited in the study using non-probability purposive sampling and were divided randomly into two equal groups; control and experimental group, by sealed envelope method. The experimental group received botulinum toxin A followed by task specific training, while the control group received only task-specific training for 12 weeks. Data was collected at baseline, after 4 weeks, 8 weeks and 12 weeks by using upper extremity items of Motor Assessment Scale and Fugl Meyer Assessment scale of upper limb, Stroke specific quality of Life, Arm dystonia Disability scale and WOLF Motor function test.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group received botulinum toxin type A. After one week of Botox administration, a specially made task specific training program was started for these patients. It was provided for a duration of one hour and for three times per week for a total of 12 weeks by a trained physiotherapist.
  Interventions: Other: Botulinum toxin type A; Other: Task Specific Training
- Control Group (Placebo Comparator): The control group received only task specific training program with the same protocol as for the experimental group; for a duration of one hour and for three times per week up to a total of 12 weeks by a trained physiotherapist
  Interventions: Other: Task Specific Training

INTERVENTIONS:
Other: Botulinum toxin type A — All patients in the experimental group received a BoNT-A injection. The injected total dose for individual patient in the experimental group was 100 units which is equivalent to approximately 300-500 Units of Dysport (the other type of BoNT-A available). The Botox was injected by the neurophysician intramuscularly using insulin U100 syringe and determination of muscles for injection was assessed clinically.
  Arms: Experimental Group
Other: Task Specific Training — Task specific training is the repetition of a specific task until expertise is reached. More challenging tasks are added as a means of progression

SUMMARY:
This study was conducted to assess the combine role of Physiotherapy by providing task specific trainings and Botulinum Toxin Type A in improving the functional outcomes of upper limb in post stroke patients with focal hand dystonia.

DETAILED DESCRIPTION:
Post-stroke hemiparesis, with dystonia, is a major cause of disability. Dystonia can hinder the functional activities making patient dependent on others for performance of daily living activities. Dystonia not only limits the physical activity of the patient but also affects their quality of life significantly. Various treatment protocols have been used in the literature for treatment of focal hand dystonia in the past including deep brain stimulation, kinesio taping, sensory oriented training, splinting, extracorporeal shock wave therapy and botox. Out of these Botox has gained much importance but it results only in improving the passive range of motion and has no consensus in improving the active range of motion and functional independence of the patient. The current study was planned to determine the effects of botulinum toxin type A combined with task-specific therapy, for post-stroke focal dystonia of upper limb.

ELIGIBILITY:
Inclusion Criteria:

* Patients having first episode of unilateral stroke
* At least 6 months of post stroke duration presenting with post stroke focal dystonia of the upper limb.
* No previous exposure of the affected hand of Botox.
* Reduced upper limb functions
* Both genders will be included equally.

Exclusion Criteria:

* Significant speech or cognitive impairment which impedes the ability to perform the assessment.
* Other significant upper limb impairment e.g. fracture or frozen shoulder within 6 months.
* Severe arthritis, amputation, evidence of fixed contracture, pregnancy or lactating womens.
* Other diagnosis likely to interfere with rehabilitation or outcome assessments, e.g. blind, malignancy,
* Other conditions which may contribute to upper limb spasticity, e.g. multiple sclerosis, cerebral palsy.
* Use of botulinum toxin to the upper limb in the previous 4 months.
* Contraindications to intramuscular injection.
* Contraindications /allergy to botulinum toxin type A, which include bleeding disorders, myasthenia gravis and concurrent use of aminoglycosides.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT): | 12 weeks
  It assessed specific changes in limb function by 19 items grouped in four subscales. The total score ranged from 0 to 57. The lower score indicated no movement and upper score indicated normal performance of the patient.
MOTOR ASSESSMENT SCALE (MAS) | 12 weeks
  It was a performance-based scale, based on a task-oriented approach to evaluate and assesses performance of functional tasks rather than isolated patterns of movement. All items were assessed using a 7-point scale from 0 - 6. A score of 6 indicated optimal motor behavior.
WOLF MOTOR FUNCTION TEST (WMFT) | 12 weeks
  It quantified motor ability through timed functional tasks. It used a 6-point ordinal scale with "0" = "does not attempt with the involved arm" to "5" = movement appears to be normal."
FUGL- MEYER ASSESSMENT TEST | 12 weeks
  It was a performance-based impairment index to measure motor functioning. The total score possible was from 0 - 66, with higher function showing the improved level of independence

SECONDARY OUTCOMES:
Severity Of Dystonia | 12 weeks
  The Arm Dystonia Disability Scale: The severity of dystonia was assessed using 0 (None) to 3 (Marked Difficulty in performing activity
Stroke Specific Quality Of Life | 12 weeks
  The stroke specific Quality Of Life was administered to patients which rated their Quality of life

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR